CLINICAL TRIAL: NCT01883843
Title: Efficacy of a Task-oriented Circuit Training Associated With Transcranial Direct Current Stimulation (tDCS) for Gait Improvement in Chronic Stroke Patients . A Randomized Controlled Trial
Brief Title: Efficacy of TOCT and (tDCS) for Gait Improvement in Patients With Chronic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, Physical Medicine and Rehabilitation doctor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stroke_tDCS_TOCT
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Stroke
Keywords: Chronic Stroke; tDCS; transcranial direct current stimulation; task oriented circuit training; TOCT; gait training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS + TOCT (Experimental): Every day will be given continuous stimulation duration of 15 minutes with intensity of 0.5 mA (for a current density of 60μA/cm2), generated by a constant current stimulator rechargeable batteries for 10 consecutive days after any rehabilitation treatment in the gym. Two sponge electrodes are placed, soaked in saline solution, fixed by an elastic band, the anode consists of an electrode oblong 8cm2 positioned at M1 area on the lower limb affection (following the medial sagittal axis, with the center of the electrode positioned at one centimeter laterally to the vertex) while the cathode (48cm2) is placed in the contralateral supraorbitale area as reference electrode.
  The current reaches 0.5mA and decreases with a ramp of 10 seconds.
  Interventions: Device: real tDCS + TOCT
- sham tDCS + TOCT (Active Comparator): Every day will be given a continuous low-intensity stimulation of 0.5mA (for a current density of 60μA/cm2) only for 10 seconds at the beginning and at the end of the stimulation for 10 consecutive days after any rehabilitative treatment. The mounting of electrodes for sham stimulation is the same used for the experimental group.
  Interventions: Device: sham tDCS + TOCT

INTERVENTIONS:
Device: sham tDCS + TOCT — Every day will be given a continuous low-intensity stimulation of 0.5mA (for a current density of 60μA/cm2) only for 10 seconds at the beginning and at the end of the stimulation for 10 consecutive days after any rehabilitative treatment. The mounting of electrodes for sham stimulation is the same used for the experimental group.
  Arms: sham tDCS + TOCT
Device: real tDCS + TOCT — Every day will be given continuous stimulation duration of 15 minutes with intensity of 0.5 mA (for a current density of 60μA/cm2), generated by a constant current stimulator rechargeable batteries for 10 consecutive days after any rehabilitation treatment in the gym. Two sponge electrodes are placed, soaked in saline solution, fixed by an elastic band, the anode consists of an electrode oblong 8cm2 positioned at M1 area on the lower limb affection (following the medial sagittal axis, with the center of the electrode positioned at one centimeter laterally to the vertex) while the cathode (48cm2) is placed in the contralateral supraorbitale area as reference electrode. The current reaches 0.5mA and decreases with a ramp of 10 seconds.
  Arms: real tDCS + TOCT

SUMMARY:
Stroke is one of the major causes of disability in the Western world. Initially gait is the most affected function, 80% of patients lose this ability.

Rehabilitation in stroke patients improves walking abilities in terms of gait and related gait activities, though six months after stroke many patients are significantly disabled.

Recently, a prospective study of 205 stroke patients showed that approximately 21% of patients have a significant decrease of mobility between the first and the third year after stroke. The main finding showed that inactivity was the most important factor for the mobility decline.

Evidence about effects of direct current brain stimulation on motor recovery function of lower limb are still little, some show that quadriceps strength after stimulation of damaged M1 area increased. Another study where tDCS was associated with robotic gait training did not report any effect compared to treatment alone. It is necessary to define if a different dosage of stimulation or the association of tDCS with gait training can improve walking and if further studies are required to investigate their effectiveness.

The aim of this clinical trial is to test the possibility of gait improvement through the association of tDCS with a specific task-oriented circuit training for walking abilities, balance and mobility.

DETAILED DESCRIPTION:
Inclusion criteria:

* Males and females subjects. Age > 18 years, <75 years.
* Diagnosis of first ischemic stroke > 6 months.
* Mini mental State Examination (MMSE) >24;
* Functional Ambulation Classification (FAC) higher or equal to 4

ELIGIBILITY:
Inclusion criteria:

* Males and females subjects. Age > 18 years, <75 years.
* Diagnosis of first ischemic stroke > 6 months.
* MMSE>24;
* FAC higher or equal to 4

Exclusion Criteria:

* Contraindications to tDCS: intracranial metal implants that can be stimulated, incorrectly positioned or over-heated by the electric current, presence of a history of epilepsy, frequent headaches or neck pain, implantable devices (ventriculoperitoneal shunts, pacemakers, intrathecal pumps, intracranial metal implants).
* Neurological or psychiatric pathology.
* Severe cardio-pulmonary, renal, hepatic diseases.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in walking abilities, balance and mobility in Six minutes walking test (6MWT) | 1)A week prior to treatment beginning 2) the week after treatment end 3) three months follow up.

SECONDARY OUTCOMES:
10 meter walking test (test of 10m) | 1)A week prior to treatment beginning 2) the week after treatment end 3)three months follow up
  walking speed test
Timed "up and go" test (TUG) | 1)A week prior to treatment beginning 2) the week after treatment end 3)three months follow up.
Unified Balance Scale (UBS) | 1)A week prior to treatment beginning 2) the week after treatment end 3)three months follow up.
Fatigue Severity Scale (FSS) | 1)A week prior to treatment beginning 2) the week after treatment end 3)three months follow up.
Stroke Impact Scale (SIS) version 3.0 | 1)A week prior to treatment beginning 2) the week after treatment end 3)three months follow up.
Stroke Specific Quality of Life (SS-QOL) | 1)A week prior to treatment beginning 2) the week after treatment end 3)three months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411